CLINICAL TRIAL: NCT03279653
Title: Effect of Sleeve Gastrectomy on Pancreatic Exocrine Insufficiency.
Brief Title: Pancreatic Exocrine Insufficiency After Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Fatih Basak, M.D., Umraniye Education and Research Hospital
Other Study IDs: p-exocrine-insufficiency
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Obesity, Morbid; Pancreatic Insufficiency
MeSH Terms: conditions — Obesity, Morbid; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SleeveGastrectomy: Sleeve Gastrectomy will be performed. Preoperative and Postoperative pancreatic enzyme sufficiency (with steatocrit or fecal elastase) will be compared.
  Interventions: Procedure: SleeveGastrectomy

INTERVENTIONS:
Procedure: SleeveGastrectomy — Preoperative enzyme test before and after sleeve gastrectomy. Sleeve Gastrectomy will be performed. Preoperative (in one month) and Postoperative (after 3 months) pancreatic enzyme sufficiency (with steatocrit or fecal elastase) will be compared.

SUMMARY:
Main proposed benefit of sleeve gastrectomy is loss of ghrelin secreting tissue. Some studies express that ghrelin augment pancreatic regeneration. Therefore we hypothesized that with sleeve gastrectomy it may result with pancreatic insufficiency.

DETAILED DESCRIPTION:
Mechanism of weight loss differs in bariatric surgery according to type of surgery.

With sleeve gastrectomy which has restrictive mechanism, ghrelin excretion decreases, and this condition is attributed as an additional mechanism in weight loss.

Ghrelin effects pancreatic regeneration, and loss of ghrelin may result with pancreatic insufficiency. Therefore we aimed to deteremine this association.

ELIGIBILITY:
Inclusion Criteria:

Patients underwent bariatric surgery (Sleeve gastrectomy) after concordonce with NIH criteria

Exclusion Criteria:

Additional operations to sleeve gastrectomy like duodenal switch. Other bariatric operations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are eligible for bariatric surgery with NIH criteria and American Society of Anesthesiologists (ASA)-Physical Status Classification System.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Pancreatic excorine enzyme difference | post operative 3 months
  Effect of operation on pancreatic excorine enzyme

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Basak, MD, Principal Investigator — University of Health Science, Umraniye Education and Research Hospital
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No